CLINICAL TRIAL: NCT05852132
Title: Clinical Study on Prognosis of Patients With Severe NPDR Undergoing Vitrectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fei Gao (Other)
Responsible Party: Sponsor-Investigator, Fei Gao, Assistant Investigator, Tianjin Medical University Eye Hospital
Organization: Tianjin Medical University Eye Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TianjinMUEHlxr0001
Record Dates: First submitted 2023-04-26; First posted 2023-05-10 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Non Proliferative Diabetic Retinopathy(NPDR)

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PPV+PRP (Experimental): PPV was performed for severe non-proliferative diabetic retinopathy with PRP.
  Interventions: Procedure: Pars plana vitrectomy(PPV) +Panretinal photocoagulation(PRP)
- Pars plana vitrectomy(PPV) (Active Comparator): Vitrectomy was performed for severe non-proliferative diabetic retinopathy, but panretinal photocoagulation(PRP) was not performed
  Interventions: Procedure: pars plana vitrectomy(PPV)
- Panretinal photocoagulation(PRP) (Placebo Comparator): Only PRP was used for severe non-proliferative diabetic retinopathy.
  Interventions: Procedure: Panretinal photocoagulation(PRP)

INTERVENTIONS:
Procedure: pars plana vitrectomy(PPV) — Vitrectomy was performed for severe non-proliferative diabetic retinopathy, but panretinal photocoagulation(PRP) was not performed
  Arms: Pars plana vitrectomy(PPV)
Procedure: Pars plana vitrectomy(PPV) +Panretinal photocoagulation(PRP) — PPV was performed for severe non-proliferative diabetic retinopathy with PRP.
  Arms: PPV+PRP
Procedure: Panretinal photocoagulation(PRP) — Only PRP was used for severe non-proliferative diabetic retinopathy.
  Arms: Panretinal photocoagulation(PRP)

SUMMARY:
To investigate the prognosis of retinal structure and function after vitrectomy in patients with severe non-proliferative diabetic retinopathy, to explore the feasibility of vitrectomy in patients with severe non-proliferative diabetic retinopathy(NPDR), and to seek the best way to delay the progression of diabetic retinopathy from the perspective of therapeutic effect.

DETAILED DESCRIPTION:
Patients were randomized into three groups according to the random number table: vitrectomy group, vitrectomy + panretinal photocoagulation group and panretinal photocoagulation group alone. 1. Vitrectomy group: vitrectomy was performed for severe non-proliferative diabetic retinopathy, but retinal laser photocoagulation was not performed. 2. Vitrectomy + panretinal photocoagulation group: vitrectomy was performed for severe non-proliferative diabetic retinopathy, and retinal laser photocoagulation was performed during the operation. 3. panretinal photocoagulation group: only retinal laser photocoagulation treatment was performed for severe non-proliferative diabetic retinopathy. All patients were regularly reviewed after surgery (preoperative, 1 week, 1 month, 3 months, 6 months, 12 months, 24 months, and the time and frequency of follow-up were increased according to the specific condition recovery), and the same physician assessed the retinal restoration and visual acuity recovery, and the follow-up time was not less than 12 months. The main outcome measures included the incidence of PDR, such as vitreous hemorrhage, the presence of neovascularization, fibroproliferative membranes, or traction retinal detachment. Secondary study endpoints included: (1) optimal corrected visual acuity; (2) Changes in the thickness of each retina layer; (3) Visual field changes; (4) area of retina without perfusion; (5) retinal neovascularization area; (6) the epiretinal membrane; (7) Low intraocular pressure/increased intraocular pressure, iris neovascularization and lens opacity, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years, men or women
2. Severe nonproliferative diabetic retinopathy was diagnosed with any one of the following, according to the International Classification of Clinical Severity of Diabetic Retinopathy: more than 20 intraretinal hemorrhaged spots in any one of four quadrants, definite venous beading in more than two quadrants, or definite intraretinal microvascular changes in more than one quadrant.
3. ETDRS beat corrected visual acuity(BCVA) letter score between 19 and 78 (Snellen equivalent 20/400-20/32) on the day of randomisation.
4. At least partial corneal transparency (or central corneal transparency), good pupil dilation and full cooperation with PRP, and ensure that the fundus examination, visual function examination and optical coherence tomography (OCT) examination can be performed after vitrectomy.
5. Able and willing to sign informed consent

Exclusion Criteria:

1. Unwilling or unable to provide consent for participation in the study, unwilling to submit to the randomisation process or unable to return for the scheduled protocol visits
2. Participating in another clinical trial within the past 3 months.
3. Previous intraocular laser therapy, intraocular surgery (excluding cataract surgery), or scheduled to undergo surgery within the next 6 months
4. Previous poorly controlled glaucoma (defined as intraocular pressure ≥25mmHg after anti-glaucoma medication)
5. Patients previously diagnosed with wet AMD, retinal vein occlusion and other neovascular retinopathy
6. Patients previously diagnosed with macular membrane, ischemic optic neuropathy, uveitis and other definite fundus diseases.
7. Received pro-VEGF or anti-VEGF treatment within the past 3 months (systemic or intravitreal).
8. Has a history of corticosteroid treatment (peribulbar or intravitreal) in the past 3 months
9. Underwent yttrium aluminum garnet capsulotomy within the past 3 months
10. Patients with intraocular fillings of silicone oil or inert gas after treatment
11. Has substantial cataract that, according to the investigator's judgement, is likely to decrease visual acuity by more than three lines (ie, the cataract reduces the visual acuity to 20/40 or worse).
12. Aphakic eye
13. Has severe external ocular infection, including conjunctivitis and substantial blepharitis.
14. Patients with severe cardiopulmonary, liver and kidney impairment and advanced cancer
15. Has blood pressure >180/110 mm Hg. If blood pressure is maintained below 180/110 mm Hg with antihypertensive medication, the individual is eligible to participate
16. Has a history of transient ischaemic attack, stroke, myocardial infarction, acute congestive heart failure or other acute cardiac event requiring hospitalization within the past 3 months.
17. For women of childbearing age: potential study participants would be questioned about pregnant, lactating or intending to become pregnant within the next 3 years. The investigator would determine when a pregnancy test is required.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 249 (Estimated)
Dates: Start 2024-05-05 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of proliferative diabetic retinopathy (PDR) | 24months postoperatively
  fluorescence fundus angiography and fundus photos are used to evaluate the fundus vessels.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin medical university eye hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No